CLINICAL TRIAL: NCT03817775
Title: Effect of Music on the Reduction of the Sedative Dose During Coronary Angioplasty: A Control-case Comparison Clinical Study
Brief Title: Effect of Music on the Sedative Use During Coronary Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Musicothérapie Applications et Recherches Cliniques (Other)
Collaborators: American Hospital of Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MusicSeda
Record Dates: First submitted 2019-01-12; First posted 2019-01-25 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Coronary Angioplasty
Keywords: Music therapy; sedation; coronary angioplasty
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from the coronary angiography patient pool of the American Hospital of Paris and assigned to one of 2 groups in a non-randomized manner: Control or music intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will undergo coronary angiography without music intervention.
- Music therapy (Experimental): The intervention group will also undergo coronary angiography and will administer music therapy between 10 minutes prior to the beginning of the procedure until its end.
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — The intervention group will administer "U" sequence between 10 minutes prior to the beginning of the procedure until its end.
  Arms: Music therapy

SUMMARY:
This is a non-blinded, non-randomized controlled pilot study with no follow-up. Patients will be recruited from the coronary angiography patient pool of the American Hospital of Paris and assigned to one of 2 groups in a non-randomized manner.

DETAILED DESCRIPTION:
This is a non-blinded, non-randomized controlled pilot study with patients who will be followed during their coronary angiography procedure and with no follow-up. Patients will be recruited from the coronary angiography patient pool of the American Hospital of Paris and assigned to one of 2 groups in a non-randomized manner. It is expected to enroll around 100 patients and this is estimated to be obtained in a period of 2 months approximately. Patients will be placed in the control group, without music intervention, or assigned to the music group. Assignment will be done in this manner due to limited availability of the hardware and software to the investigation team. Patients in both groups will be matched based on age, sex, weight, height, American Society of Anesthesiology (ASA) score, and prior medical history, including diabetes, hypertension, chronic kidney disease and stroke. Each patient will receive a standardized sedation in the traditional manner and at the discretion of the investigator to reach Bispectral index (BIS) score below 90 and sedation score ≤ 1. The primary study end points will be the consumptions in analgesics and hypnotics. Secondary study end points will be pain and anxiety scores as measured the Numeric Rating Scale (NRS), the Visual Analog Scale (VAS) and the Amsterdam Preoperative Anxiety and Information Scale (APAIS).

ELIGIBILITY:
Inclusion Criteria:

* Patient needs a coronary angiography
* Patient gives verbal consent to participation in the study.

Exclusion Criteria:

* Patient aged less than 18 years at time of enrollment
* Patient doesn't like music for cultural reason
* Patient with serious psychiatric disorders
* Patient with not paired deafness or paired one with devices that are incompatible with wearing a headset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BOCCARA, PhD, Principal Investigator — Department of Anaesthesia and Intensive Care, American Hospital of Paris
Locations (1):
- American Hospital of Paris, Neuilly-sur-Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaber S, Bahloul H, Guetin S, Chanques G, Sebbane M, Eledjam JJ. [Effects of music therapy in intensive care unit without sedation in weaning patients versus non-ventilated patients]. Ann Fr Anesth Reanim. 2007 Jan;26(1):30-8. doi: 10.1016/j.annfar.2006.09.002. Epub 2006 Nov 3. French. PMID 17085009
- [Background] Guetin S, Ginies P, Siou DK, Picot MC, Pommie C, Guldner E, Gosp AM, Ostyn K, Coudeyre E, Touchon J. The effects of music intervention in the management of chronic pain: a single-blind, randomized, controlled trial. Clin J Pain. 2012 May;28(4):329-37. doi: 10.1097/AJP.0b013e31822be973. PMID 22001666
- [Background] Messika J, Hajage D, Panneckoucke N, Villard S, Martin Y, Renard E, Blivet A, Reignier J, Maquigneau N, Stoclin A, Puechberty C, Guetin S, Dechanet A, Fauquembergue A, Gaudry S, Dreyfuss D, Ricard JD. Effect of a musical intervention on tolerance and efficacy of non-invasive ventilation in the ICU: study protocol for a randomized controlled trial (MUSique pour l'Insuffisance Respiratoire Aigue - Mus-IRA). Trials. 2016 Sep 13;17(1):450. doi: 10.1186/s13063-016-1574-z. PMID 27618935
- [Background] Guetin S, Brun L, Deniaud M, Clerc JM, Thayer JF, Koenig J. Smartphone-based Music Listening to Reduce Pain and Anxiety Before Coronarography: A Focus on Sex Differences. Altern Ther Health Med. 2016 Jul;22(4):60-3. PMID 27548494

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: The control group underwent coronary angiography without music intervention.
- Music Therapy: The intervention group also underwent coronary angiography and administered music therapy between 10 minutes prior to the beginning of the procedure until its end.
  Music therapy: The intervention group administered "U" sequence between 10 minutes prior to the beginning of the procedure until its end.
Period: Overall Study
Arm/Group | Control | Music Therapy
Started | 22 | 54
Completed | 22 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Music Therapy | Total
Number analyzed (Participants) | 22 | 54 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (13.37) | 67.2 (9.07) | 65.7 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 18 | 48 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 22 | 54 | 76
ASA Score [Count of Participants; unit: Participants]
  Normal: Score 1 | 2 | 0 | 2
  Moderate abnormality: Score 2 | 3 | 5 | 8
  Severe abnormality: Score 3 | 16 | 45 | 61
  Missing | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose Use of Midazolam Medication (mg)
Description: The consumption in Midazolam medication was reported during the coronary angioplasty. Dose was in mg.
Time Frame: Between 10 minutes prior to the beginning of the procedure up to 45 minutes.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 22 | 54
mg | 3.0 (0.84) | 1.2 (0.76)
Statistical Analysis 1: Comparison: Control vs Music Therapy; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Dose Use of Propofol Medication (mg)
Description: The consumption in Propofol medication was reported during the coronary angioplasty. Dose was in mg.
Time Frame: Between 10 minutes prior to the beginning of the procedure up to 45 minutes.
Population: One patient in control group and 2 patients in music therapy group had missing data on Propofol medication.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 21 | 52
mg | 12.8 (21.83) | 52 (0)
Statistical Analysis 1: Comparison: Control vs Music Therapy; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Dose Use of Sufentanil Medication (ug)
Description: The consumption in Sufentanil medication was reported during the coronary angioplasty. Dose was in ug.
Time Frame: Between 10 minutes prior to the beginning of the procedure up to 45 minutes.
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 22 | 54
ug | 4.9 (1.21) | 5.1 (1.02)
Statistical Analysis 1: Comparison: Control vs Music Therapy; Test type: Other; p = 0.7215, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Pain Score
Description: Pain score was measured using the Visual Analog Scale (VAS). This scale ranged from 0 (no pain) to 10 (very high pain), and collected the maximum pain the patient had during the procedure. This was collected right after the end of the procedure in the recovery room.
Time Frame: From 0 up to 45 minutes.
Population: Three patients in control group and 3 patients in music therapy group had missing data on VAS pain score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 19 | 51
score on a scale | 0.5 (0.70) | 0.7 (1.47)
Statistical Analysis 1: Comparison: Control vs Music Therapy; Test type: Other; p = 0.5675, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Anxiety Score (NRS)
Description: Anxiety score was measured using the Numeric Rating Scale (NRS). This scale ranged from 0 (no anxiety) to 10 (very high anxiety), and collected the maximum anxiety the patient had during the procedure. This was collected right after the end of the procedure in the recovery room.
Time Frame: From 0 up to 45 minutes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 21 | 53
score on a scale | 4.2 (1.89) | 2.9 (2.19)
Statistical Analysis 1: Comparison: Control vs Music Therapy; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Satisfaction of the Patient
Description: Satisfaction was measured using a scale from 0 to 5, with a higher score for a high satisfaction.
Time Frame: Right after the end of the procedure in the recovery room.
Population: Two patients in control group and 3 patients in music therapy group had missing data on satisfaction endpoint.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 20 | 51
Score | 4.5 (0.51) | 4.8 (0.44)

7. Secondary Outcome: Effect on Physiological Parameters: BIS
Description: Bispectral index (BIS) score at baseline which corresponds to 10 minutes before the beginning of the procedure.
  The BIS monitor provides a single dimensionless number which ranges from 0 (equivalent to EEG silence) to 100. Higher is the score, better it is.
Time Frame: 10 minutes prior to the beginning of the procedure
Population: 2 missing data in control group
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 20 | 54
Score | 96.9 (2.1) | 94.9 (5.5)

8. Secondary Outcome: Effect on Physiological Parameters: Heart Rate
Description: Heart rate at Baseline which corresponds to 10 minutes before the beginning of the procedure.
Time Frame: 10 minutes prior to the beginning of the procedure.
Measure: Mean (Standard Deviation); unit: beat/min
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 22 | 54
beat/min | 71.3 (13.1) | 65.5 (11.4)

9. Secondary Outcome: Effect on Physiological Parameters: SpO2%
Description: SpO2 at Baseline which corresponds to 10 minutes before the beginning of the procedure..
Time Frame: 10 minutes prior to the beginning of the procedure.
Measure: Mean (Standard Deviation); unit: Percentage of O2 saturation in blood
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 22 | 54
Percentage of O2 saturation in blood | 98.5 (1.4) | 98.9 (1.3)

10. Secondary Outcome: Effect on Physiological Parameters: Mean Arterial Blood Pressure
Description: Mean arterial blood pressure at Baseline which corresponds to 10 minutes before the beginning of the procedure.
Time Frame: 10 minutes prior to the beginning of the procedure.
Population: Two patients in control group and 1 in music therapy had missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 20 | 53
mmHg | 104.7 (14.1) | 104.2 (17.2)

ADVERSE EVENTS:
Time Frame: From 0 up to 45 minutes
Arm/Group | Control | Music Therapy
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/54
Other Adverse Events (participants affected / at risk) | 0/22 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03817775/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT03817775/SAP_001.pdf